CLINICAL TRIAL: NCT03288688
Title: Effect of an Exercise Program Designed for Professional Orchestral Musicians on Performance-related Musculoskeletal Problems - a Randomized Controlled Trial
Brief Title: Effect of an Exercise Program Designed for Orchestral Musicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Jean-Sébastien Roy, PhD, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Orch musicians
Record Dates: First submitted 2017-09-18; First posted 2017-09-20 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Musculoskeletal Disorder
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise program and education (Experimental): An exercise program in the form of home exercise videos will be given to the participants in this group. They will be asked to perform a minimum of two 35-minute exercise sessions per week, over a period of 11 weeks. They will also be required to attend three group exercise sessions, to confirm correct execution of the exercises. A short educational presentation on injury prevention will be offered at the beginning of the study, followed by three informative e-mails over the course of the study.
  Interventions: Other: Exercise program and education
- No intervention (No Intervention): Participants in this group will be asked to continue their usual activities.

INTERVENTIONS:
Other: Exercise program and education — The exercise program comprises warm-ups, exercises and cool-downs and aims to improve recruitment, strength and endurance of postural muscle groups that are key to the work of a musician. Basic activation exercises progress to dynamic and resisted exercises as well as functional musical movements. There is a series of six exercises of increasing difficulty for each of the following bodily regions: hips, back, neck, shoulders and abdominals.
  Topics to be discussed in the educational presentation and e-mails include healthy practice habits, activity dosage, the importance of physical activity, how the body adapts to workload and physical stressors, and instructions pertaining to the exercise program.
  Arms: Exercise program and education

SUMMARY:
This study is a randomized clinical trial evaluating the effect of an exercise program designed specifically for orchestral musicians on performance-related musculoskeletal problems (PRMPs). Professional and conservatory-level orchestral musicians will be recruited. Half of the subjects will participate in an 11-week home exercise program and attend three group exercise sessions and an educational presentation on injury prevention, while the other half of the subjects will receive no intervention, and continue their usual activities.

ELIGIBILITY:
Inclusion Criteria:

* professional or freelance orchestral musician, or tertiary-level full-time music student majoring in an orchestral instrument
* able to commit to performing exercises 2 times per week over an 11-week period
* medical condition permitting participation in an exercise program (ie. no serious heart or lung condition that may be exacerbated by physical exertion)

Exclusion Criteria:

* presence of musculoskeletal injuries definitively non-related to musical practice or performance
* fewer than 15 hours per week playing their instrument
* corticosteroid infiltration in the 6 weeks preceding recruitment
* prescribed anti-inflammatory drugs or neurontin in the 3 weeks preceding recruitment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2017-11-17 (Actual); Study Completion 2017-11-17 (Actual)

PRIMARY OUTCOMES:
The Musculoskeletal Pain Intensity and Interference Questionnaire for professional orchestra Musicians (MPIIQM) | Baseline-11 weeks
  A biopsychosocial self-report questionnaire used to obtain demographic and occupational information and to document the intensity and impact of performance-related musculoskeletal pain/problems

SECONDARY OUTCOMES:
The Nordic Musculoskeletal Questionnaire (NMQ) | Baseline-11 weeks
  Self-report questionnaire on pain/symptom prevalence in the different regions of the body
Global Rating of Change | 11 weeks
  Questionnaire designed to quantify participants' perceived improvement or deterioration over the course of the study

CONTACTS AND LOCATIONS:
Locations (1):
- CIRRIS, Québec, Quebec, Canada